CLINICAL TRIAL: NCT03654274
Title: SPIRIT EXTENSION: An International Phase 3 Open-Label, Single-Arm, Safety and Efficacy Extension Study to Evaluate Relugolix Co-Administered With Low-Dose Estradiol and Norethindrone Acetate in Women With Endometriosis-Associated Pain
Brief Title: SPIRIT EXTENSION: Efficacy and Safety Extension Study of Relugolix in Women With Endometriosis-Associated Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601-3103; 2017-004066-10 (EudraCT Number)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; Dysmenorrhea; Pain; Dyspareunia; Pelvic Pain
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Pain; Dyspareunia; Pelvic Pain | interventions — relugolix; estradiol, norethindrone drug combination

STUDY DESIGN:
Intervention Model Description: Open label extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relugolix plus E2/NETA (Experimental): Relugolix co-administered with E2/NETA for 80 weeks.
  Interventions: Drug: Relugolix; Drug: Estradiol/norethindrone acetate

INTERVENTIONS:
Drug: Relugolix — Relugolix 40-mg tablet administered orally once daily
  Other Names: TAK-385; MVT-601
Drug: Estradiol/norethindrone acetate — Capsule containing co-formulated tablet of E2 (1.0 mg) and NETA (0.5 mg) administered orally once daily
  Other Names: E2/NETA; low-dose hormonal add-back

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety of relugolix 40 milligram (mg) once daily co-administered with low-dose estradiol (E2) and norethindrone acetate (NETA) for up to 104 weeks on endometriosis-associated pain in participants who previously completed a 24-week treatment period in one of the parent studies (MVT-601-3101 or MVT-601-3102).

DETAILED DESCRIPTION:
This study is an international phase 3 open-label, single-arm, long-term efficacy and safety extension study that will enroll eligible participants who have completed their participation in one of the phase 3 randomized, double-blind, placebo-controlled parent studies, MVT-601-3101 (SPIRIT 1 - NCT03204318) or MVT-601-3102 (SPIRIT 2 - NCT03204331). All participants will receive relugolix 40 mg orally once daily co-administered with low-dose E2 (1.0 mg) and NETA (0.5 mg) for 80 weeks.

Approximately 800 women with endometriosis-associated pain will be enrolled, after having completed a 24-week treatment period in one of the parent studies. The objectives of the study are to evaluate long-term efficacy and safety through up to 104 weeks of treatment (including treatment during the parent study) of relugolix co-administered with low-dose E2/NETA.

Baseline procedures for this extension study will be performed on the same day as the Week 24 Visit of the parent study. This visit, referred to as the "Week 24/Baseline Visit, will be defined as the date of completion of the last Week 24 procedure in the parent study. Participants will have received their last dose of study drug in the parent study on the day prior to the Week 24/Baseline Visit and will receive their first dose of study drug for this extension study in the clinic after the participant is determined to be eligible for this extension study and has provided informed consent to participate. The administration of the first dose of study drug for MVT-601-3103 will define enrollment into this study. Study participants will then take the open-label study treatment orally, once daily for 80 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Completed 24 weeks of study drug treatment and study participation in either parent study, MVT-601-3101 or MVT-601-3102.
2. Is not expected to undergo gynecological surgery or other surgical procedures for treatment of endometriosis (including ablation, shaving, or excision) during the study, including during the Follow-Up Period, and the participant does not desire such treatment during this time frame.
3. Has agreed to continue to use only study-specified analgesic medications during the study and is not known to be intolerant to these.

Key Exclusion Criteria:

1. Has had a surgical procedure for treatment for endometriosis at any time during the parent study (MVT-601-3101 or MVT-601-3102).
2. Has any chronic pain or frequently recurring pain condition, other than endometriosis, that is treated with opioids or requires analgesics for ≥ 7 days per month.
3. Has a Z-score < -2.0 or has a ≥ 7% decrease in bone mineral density from the parent study Baseline at lumbar spine, total hip, or femoral neck based on the parent study Week 24 DXA assessment of bone mineral density.
4. Has any contraindication to treatment with low-dose E2 and NETA, including:

   1. Known, suspected, or history of breast cancer;
   2. Known or suspected estrogen-dependent neoplasia;
   3. Active deep vein thrombosis or pulmonary embolism, or history of these conditions prior to the Week 24/Baseline visit;
   4. History of or active arterial thromboembolic disease, including stroke and myocardial infarction;
   5. Known anaphylactic reaction or angioedema or hypersensitivity to E2 or NETA;
   6. Known protein C, protein S, or antithrombin deficiency, or other known thrombophilia disorders, including Factor V Leiden;
   7. Migraine with aura;
   8. History of porphyria.
5. Had any of the following clinical laboratory abnormalities at the parent study Week 20 visit or, if available, any subsequent visit in one of the parent studies (MVT-601-3101 or MVT-601-3102):

   1. Alanine aminotransferase or aspartate aminotransferase > 2.0 times the upper limit of normal (ULN); or
   2. Bilirubin (total bilirubin) > 1.5 x ULN (or > 2.0 x ULN if secondary to Gilbert syndrome or pattern consistent with Gilbert syndrome).

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 802 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myovant Medical Monitor, Study Director — Myovant Sciences
Locations (140):
- United States (54):
  - Andalusia, Andalusia, Alabama
  - Scottsdale, Scottsdale, Arizona
  - Tucson, Tucson, Arizona
  - Tuscon, Tucson, Arizona
  - Canoga Park, Canoga Park, California
  - Los Angeles, Los Angeles, California
  - San Diego, San Diego, California
  - Greenwood Village, Greenwood Village, Colorado
  - Washington, Washington D.C., District of Columbia
  - Aventura, Aventura, Florida
  - Fort Myers, Fort Myers, Florida
  - Hialeah, Hialeah, Florida
  - Margate, Margate, Florida
  - Miami, Miami, Florida
  - Sarasota, Sarasota, Florida
  - Tampa, Tampa, Florida
  - Atlanta, Atlanta, Georgia
  - Augusta, Augusta, Georgia
  - Norcross, Norcross, Georgia
  - Idaho Falls, Idaho Falls, Idaho
  - Oakbrook, Oakbrook Terrace, Illinois
  - Park Ridge, Park Ridge, Illinois
  - Shawnee, Shawnee Mission, Kansas
  - Marrero, Marrero, Louisiana
  - Towson, Towson, Maryland
  - Saginaw, Saginaw, Michigan
  - Jefferson City, Jefferson City, Missouri
  - St. Louis, St Louis, Missouri
  - Omaha, Omaha, Nebraska
  - Las Vegas, Las Vegas, Nevada
  - Durham, Durham, North Carolina
  - New Bern, New Bern, North Carolina
  - Winston Salem, Winston-Salem, North Carolina
  - Akron, Akron, Ohio
  - Columbus, Columbus, Ohio
  - Englewood, Englewood, Ohio
  - Hershey, Hershey, Pennsylvania
  - Columbia, Columbia, South Carolina
  - Chattanooga, Chattanooga, Tennessee
  - Memphis, Memphis, Tennessee
  - Beaumont, Beaumont, Texas
  - Corpus Christi, Corpus Christi, Texas
  - Dallas, Dallas, Texas
  - Fort Worth, Fort Worth, Texas
  - Houston, Houston, Texas
  - Irving, Irving, Texas
  - San Antonio, San Antonio, Texas
  - Sugar Land, Sugar Land, Texas
  - Webster, Webster, Texas
  - Salt Lake City, Salt Lake City, Utah
  - Norfolk, Norfolk, Virginia
  - Richmond, Richmond, Virginia
  - Virginia Beach, Virginia Beach, Virginia
  - Seattle, Seattle, Washington
- Argentina (4):
  - Ciudad de Buenos Aires, Ciudad de Buenos Aires, Buenos Aires
  - San Isidro, San Isidro, Buenos Aires
  - Rosario, Rosario, Santa Fe Province
  - Cordoba, Córdoba
- Australia (5):
  - Sydney, Sydney, New South Wales
  - Wollongong, Wollongong, NS
  - Taringa, Taringa, Queensland
  - Adelaide, Adelaide, South Australia
  - Nedlands, Nedlands, Western Australia
- Belgium (4):
  - Leuven, Leuven, Flemish Brabant
  - La Louvière, La Louvière, Hainaut
  - Gent, Ghent, Oost-vlaanderen
  - Brussels, Brussels
- Brazil (7):
  - Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Porto Alegre, Porto Alegre, São Paulo
  - São Bernardo do Campo, São Bernardo do Campo, São Paulo
  - São Paulo, São Paulo, São Paulo
  - Sao Paulo, São Paulo, São Paulo
  - Sao Paulo, São Paulo
- Bulgaria (5):
  - Sofia, Sofia, Sofia
  - Blagoevgrad, Blagoevgrad
  - Pleven, Pleven
  - Stara Zagora, Stara Zagora
  - Varna, Varna
- Canada (3):
  - Red Deer, Red Deer, Alberta
  - Waterloo, Waterloo, Ontario
  - Victoriaville, Victoriaville, Quebec
- Santiago, Santiago, Chile
- Czechia (9):
  - Tábor, Tábor, Jihormoravsky Kraj
  - Písek, Písek, Jihočeský kraj
  - Vodňany, Vodňany, Jihočeský kraj
  - Náchod, Náchod, Královéhradecký kraj
  - Praha 10, Prague, Prague
  - Praha 2, Prague, Prague
  - České Budějovice, České Budějovice
  - Olomouc, Olomouc
  - Praha 8 - Libeň, Praha 8 - Libeň
- Finland (3):
  - Kuopio, Kuopio, Eastern Finland
  - Helsinki, Helsinki, Southern Finland
  - Oulu, Oulu
- Tbilisi, Tbilisi, Georgia
- Hungary (7):
  - Pécs, Pécs, Baranya
  - Békéscsaba, Békéscsaba, Bekes County
  - Gyula, Gyula, Bekes County
  - Kecskemét, Kecskemét, Bács-Kiskun county
  - Szeged, Szeged, Csongrád megye
  - Debrecen, Debrecen, Hajdú-Bihar
  - Nyíregyháza, Nyíregyháza, Szabolcs-Szatmár-Bereg
- Italy (5):
  - Monserrato, Monserrato, Cagliari
  - Catanzaro, Catanzaro
  - Napoli, Napoli
  - Pavia, Pavia
  - Roma, Roma
- New Zealand (3):
  - Remuera, Remuera, Auckland
  - Palmerston North, Palmerston North, Manawatu-Wanganui
  - Christchurch, Christchurch
- Poland (7):
  - Skórzewo, Skórzewo, Greater Poland Voivodeship
  - Lublin, Lublin, Lublin Voivodeship
  - Warszawa, Warsaw, Masovian Voivodeship
  - Białystok, Bialystok, Podlaskie Voivodeship
  - Katowice, Katowice, Silesian Voivodeship
  - Szczecin, Szczecin, West Pomeranian Voivodeship
  - Łódź, Lodz, Łódź Voivodeship
- Portugal (4):
  - Almada, Almada, Lisbon District
  - Coimbra, Coimbra
  - Covilhã, Covilha
  - Porto, Porto
- Romania (3):
  - Brasov, Brasov
  - Bucuresti, Bucharest
  - București, Bucharest
- South Africa (5):
  - Port Elizabeth, Port Elizabeth, Eastern Cape
  - Centurion, Centurion, Gauteng
  - Roodepoort, Roodepoort, Gauteng
  - Durban, Durban, KwaZulu-Natal
  - Cape Town, Cape Town, Western Cape
- Spain (2):
  - Madrid, Madrid
  - Valencia, Valencia
- Ukraine (8):
  - Kyiv, Kyiv, Kiev City
  - Kyiv, Kyiv, Kyiv City
  - Chernivtsi, Chernivtsi
  - Ivano-Frankivsk, Ivano-Frankivsk
  - Kharkiv, Kharkiv
  - Kiev, Kiev
  - Kyiv, Kyiv
  - Zaporizhzhya, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] As-Sanie S, Abrao MS, Reznichenko G, Wilk K, Zhong Y, Perry J, Hunsche E, Soulban G, Becker CM. Impact of relugolix combination therapy on functioning and quality of life in women with endometriosis-associated pain. Fertil Steril. 2024 Oct;122(4):687-695. doi: 10.1016/j.fertnstert.2024.06.009. Epub 2024 Jun 19. PMID 38906210
- [Derived] Becker CM, Johnson NP, As-Sanie S, Arjona Ferreira JC, Abrao MS, Wilk K, Imm SJ, Mathur V, Perry JS, Wagman RB, Giudice LC. Two-year efficacy and safety of relugolix combination therapy in women with endometriosis-associated pain: SPIRIT open-label extension study. Hum Reprod. 2024 Mar 1;39(3):526-537. doi: 10.1093/humrep/dead263. PMID 38243752

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who completed their participation in one of the pivotal studies (MVT-601-3101 or MVT-601-3102) were eligible to enroll in this study.
Pre-assignment Details: The study results were presented by pivotal study treatment but all the participants only received relugolix plus Estradiol (E2)/Norethindrone Acetate (NETA).
Groups:
- Relugolix Plus E2/NETA (Group A): Relugolix 40 mg once daily co-administered with E2 (1 mg) and NETA (0.5 mg) for 24 weeks in the pivotal study followed by Relugolix 40 mg once daily co-administered with E2/NETA for 80 weeks in this extension study.
- Relugolix Plus Delayed E2/NETA (Group B): Relugolix 40 mg monotherapy (once daily) for 12 weeks, followed by oral relugolix 40 mg once daily co-administered with E2 (1mg) and NETA (0.5 mg) for 12 weeks in the pivotal study and Relugolix 40 mg once daily co-administered with E2/NETA for 80 weeks in this extension study.
- Placebo (Group C): Relugolix placebo co-administered with E2/NETA placebo for up to 24 weeks in the pivotal study followed by Relugolix 40 mg once daily co-administered with E2/NETA for 80 weeks in this extension study.
Period: Overall Study
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Started | 278 | 247 | 277
Received at Least 1 Dose of Study Drug | 277 | 247 | 275
Completed | 172 | 155 | 174
Not Completed | 106 | 92 | 103
Not completed — Adverse Event | 19 | 23 | 24
Not completed — Protocol Deviation | 0 | 2 | 0
Not completed — Lost to Follow-up | 8 | 6 | 5
Not completed — Withdrawal by Subject | 46 | 25 | 33
Not completed — Lack of Efficacy | 4 | 5 | 7
Not completed — Pregnancy | 2 | 2 | 1
Not completed — Other | 27 | 29 | 32
Not completed — Participants Who Consented to Week 52 and Completed at Week 52 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Extension Study Population: all participants who enrolled into MVT-601-3103 study and received any amount of open-label study drug in MVT-601-3103 study. Three participants (1 in the relugolix plus E2/NETA group and 2 in the placebo group) were excluded due to Good Clinical Practice noncompliance at Site 3015 and no data is reported for these patients. Study results are reported by pivotal study treatment, but all participants only received relugolix plus E2/NETA.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C) | Total
Number analyzed (Participants) | 277 | 247 | 275 | 799
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 277 | 247 | 275 | 799
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 247 | 275 | 799
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 31 | 42 | 100
  Not Hispanic or Latino | 249 | 215 | 233 | 697
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Number of participants based on their race.
  Participants
    American Indian or Alaska Native | 1 | 1 | 0 | 2
    Asian | 0 | 1 | 0 | 1
    Black or African American | 17 | 7 | 13 | 37
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
    White | 254 | 236 | 248 | 738
    Other | 1 | 0 | 8 | 9
    Multiple | 4 | 2 | 5 | 11
    Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 44 | 52 | 144
  Argentina | 10 | 12 | 12 | 34
  Australia | 2 | 4 | 5 | 11
  Belgium | 3 | 2 | 3 | 8
  Brazil | 13 | 13 | 15 | 41
  Bulgaria | 14 | 5 | 10 | 29
  Canada | 0 | 2 | 4 | 6
  Chile | 3 | 1 | 1 | 5
  Czechia | 12 | 8 | 8 | 28
  Finland | 2 | 2 | 1 | 5
  Georgia | 5 | 1 | 1 | 7
  Hungary | 7 | 10 | 7 | 24
  Italy | 7 | 8 | 2 | 17
  New Zealand | 2 | 2 | 4 | 8
  Poland | 105 | 86 | 106 | 297
  Portugal | 1 | 4 | 2 | 7
  Romania | 12 | 12 | 7 | 31
  South Africa | 8 | 10 | 14 | 32
  Spain | 0 | 1 | 1 | 2
  Ukraine | 23 | 20 | 20 | 63
Time Since Surgical Diagnosis of Endometriosis [Mean (Standard Deviation); unit: years] | 4.0 (3.52) | 4.7 (4.00) | 3.9 (3.24) | 4.2 (3.60)
Dysmenorrhea Numerical Rating Scale (NRS) Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Assessed using an NRS score (11-point scale) for pain recorded daily in an electronic diary. Higher NRS score means worse condition (0 = no pain to 10 = pain as bad as you can imagine).
  score on a scale | 7.1 (1.66) | 7.0 (1.65) | 7.2 (1.63) | 7.1 (1.65)
Nonmenstrual Pelvic Pain (NMPP) NRS Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Assessed using an NRS score (11-point scale) for pain recorded daily in an electronic diary. Higher NRS score means worse condition (0 = no pain to 10 = pain as bad as you can imagine).
  score on a scale | 5.7 (1.93) | 5.5 (1.98) | 5.7 (1.91) | 5.6 (1.94)
Bone Mineral Density (BMD) Lumbar Spine L1-L4 [Mean (Standard Deviation); unit: g/cm^2] | 1.14 (0.163) | 1.14 (0.144) | 1.14 (0.149) | 1.14 (0.153)
BMD Total Hip [Mean (Standard Deviation); unit: g/cm^2] | 0.98 (0.133) | 0.97 (0.120) | 0.98 (0.123) | 0.97 (0.126)
BMD Femoral Neck [Mean (Standard Deviation); unit: g/cm^2] | 0.93 (0.157) | 0.92 (0.136) | 0.93 (0.151) | 0.92 (0.149)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants Who Meet The Dysmenorrhea Responder Criteria At Week 52
Description: Assessed using an NRS score (11-point scale) for pain recorded daily in an electronic diary. A participant was defined as a responder if the NRS score for dysmenorrhea declined from baseline to Week 52 by at least 2.8 points without increased use of protocol-specified analgesics for pelvic pain at Week 52 relative to baseline. Participants rated their pelvic pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating pain as bad as you can imagine.
Time Frame: Week 52
Population: Extension Study Population: all participants who enrolled into MVT-601-3103 study and received any amount of open-label study drug in MVT-601-3103 study. Study results are reported by pivotal study treatment, but all participants only received relugolix plus E2/NETA.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 277 | 247 | 275
percentage of participants | 84.8 [80.06 to 88.85] | 82.2 [76.83 to 86.75] | 75.6 [70.12 to 80.59]

2. Primary Outcome: Percentage Of Participants Who Meet The NMPP Responder Criteria At Week 52
Description: Assessed using an NRS score (11-point scale) for pain recorded daily in an electronic diary. A participant was defined as a responder if the NRS score for NMPP declined from baseline to Week 52 by at least 2.1 points without increased use of protocol-specified analgesics for pelvic pain at Week 52 relative to baseline. Participants rated their pelvic pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating pain as bad as you can imagine.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 277 | 247 | 275
percentage of participants | 73.6 [68.04 to 78.74] | 70.4 [64.33 to 76.06] | 68.0 [62.13 to 73.47]

3. Primary Outcome: Percentage Of Participants Who Meet The Dysmenorrhea Responder Criteria At Week 104
Description: Assessed using an NRS score (11-point scale) for pain recorded daily in an electronic diary. A participant was defined as a responder if the NRS score for dysmenorrhea declined from baseline to Week 104 by at least 2.8 points without increased use of protocol-specified analgesics for pelvic pain at Week 104 relative to baseline. Participants rated their pelvic pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating pain as bad as you can imagine.
Time Frame: Week 104
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 277 | 247 | 275
percentage of participants | 84.8 [80.06 to 88.85] | 83.0 [77.72 to 87.46] | 80.4 [75.17 to 84.89]

4. Primary Outcome: Percentage Of Participants Who Meet The NMPP Responder Criteria At Week 104
Description: Assessed using an NRS score (11-point scale) for pain recorded daily in an electronic diary. A participant was defined as a responder if the NRS score for NMPP declined from baseline to Week 104 by at least 2.1 points without increased use of protocol-specified analgesics for pelvic pain at Week 104 relative to baseline. Participants rated their pelvic pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating pain as bad as you can imagine.
Time Frame: Week 104
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 277 | 247 | 275
percentage of participants | 75.8 [70.33 to 80.74] | 71.7 [65.60 to 77.19] | 73.1 [67.44 to 78.24]

5. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Endometriosis Health Profile (EHP)-30 Pain Domain Scores At Week 52
Description: Assessed using the pain domain of the EHP-30 questionnaire. The EHP-30 questionnaire was completed on an electronic tablet (eTablet) device. Participants reported the frequency (never, rarely, sometimes, often, and always) with which they had difficulty with activities such as standing, sitting, walking, sleeping, and performing jobs around the house because of pain. The Pain Domain normalized scores ranged from 0 to 100, with higher scores denoting greater functional impact of pain. The least squares (LS) mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: Extension Study Population: all participants who enrolled into MVT-601-3103 study and received any amount of open-label study drug in MVT-601-3103 study. Study results are reported by pivotal study treatment, but all participants only received relugolix plus E2/NETA. The overall number of participants analyzed represents the number of participants evaluable at that time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 232 | 207 | 229
score on a scale | -37.7 (1.34) | -36.1 (1.37) | -35.1 (1.32)

6. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Endometriosis Health Profile (EHP)-30 Pain Domain Scores At Week 104
Description: as for outcome 5
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 167 | 151 | 173
score on a scale | -41.3 (1.33) | -38.9 (1.36) | -37.7 (1.29)

7. Secondary Outcome: Percentage Of Participants Who Have A Reduction Of At Least 20 Points In The EHP-30 Pain Domain Scores From The Pivotal Phase 3 Study Baseline At Week 52
Description: Assessed using the Pain Domain of the EHP-30 questionnaire. The EHP-30 questionnaire was completed on an electronic tablet (eTablet) device. Participants reported the frequency (never, rarely, sometimes, often, and always) with which they had difficulty with activities such as standing, sitting, walking, sleeping, and performing jobs around the house because of pain. The Pain Domain normalized scores ranged from 0 to 100, with higher scores denoting greater functional impact of pain.
Time Frame: Week 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Relugolix Plus Delayed E2/NETA (Group B): Relugolix 40 mg monotherapy (once daily) for 12 weeks, followed by oral relugolix 40 mg once daily co-administered with E2 (1mg) and NETA (0.5 mg) for 12 weeks in the pivotal study.
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 232 | 207 | 229
percentage of participants | 83.6 [78.22 to 88.14] | 81.2 [75.16 to 86.25] | 79.5 [73.66 to 84.51]

8. Secondary Outcome: Percentage Of Participants Who Have A Reduction Of At Least 20 Points In The EHP-30 Pain Domain Scores From The Pivotal Phase 3 Study Baseline At Week 104
Description: as for outcome 7
Time Frame: Week 104
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 167 | 151 | 173
percentage of participants | 88.6 [82.80 to 93.01] | 85.4 [78.78 to 90.64] | 86.1 [80.06 to 90.90]

9. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean Dysmenorrhea NRS Score At Week 52
Description: Assessed using an NRS score (11-point scale) for pain recorded daily in an electronic diary. Participants rated their pelvic pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating pain as bad as you can imagine. The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 235 | 204 | 233
score on a scale | -5.9 (0.15) | -5.7 (0.16) | -5.3 (0.15)

10. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean Dysmenorrhea NRS Score At Week 104
Description: as for outcome 9
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Relugolix Plus Delayed E2/NETA (Group B): Relugolix 40 mg monotherapy (once daily) for 12 weeks, followed by oral relugolix 40 mg once daily co-administered with E2 (1mg) and NETA (0.5 mg) for 12 weeks in the pivotal study, and Relugolix 40 mg once daily co-administered with E2/NETA for 80 weeks in this extension study.
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 112 | 124
score on a scale | -5.9 (0.17) | -5.7 (0.18) | -5.6 (0.17)

11. Secondary Outcome: Percentage Of Participants Who Are "Better" Or "Much Better" On The Patient Global Impression Of Change (PGIC) For Dysmenorrhea At Week 52
Description: The PGIC for dysmenorrhea is a 1-item questionnaire designed to assess participant's impression of change in the severity of pain during their menstrual cycle. The questionnaire used a 7-point response scale: much better, better, a little better, the same, a little worse, worse, or much worse.
Time Frame: Week 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 221 | 202 | 230
percentage of participants | 89.1 [84.27 to 92.92] | 87.1 [81.71 to 91.42] | 83.0 [77.56 to 87.66]

12. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean NMPP NRS Score At Week 52
Description: as for outcome 9
Time Frame: Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 235 | 204 | 233
score on a scale | -3.6 (0.15) | -3.4 (0.16) | -3.4 (0.15)

13. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean NMPP NRS Score At Week 104
Description: as for outcome 9
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 112 | 124
score on a scale | -4.0 (0.16) | -3.5 (0.17) | -3.8 (0.16)

14. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean Overall Pelvic Pain NRS Score At Week 52
Description: Assessed using an NRS score (11-point scale) for overall pain recorded daily in an electronic diary. Participants rated their overall pelvic pain on a scale from 0 to 10, with 0 indicating no pain and 10 indicating pain as bad as you can imagine. The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: Extension Study Population: all participants who enrolled into MVT-601-3103 study and received any amount of open-label study drug in MVT-601-3103 study. Study results are reported by pivotal study treatment, but all participants only received relugolix plus E2/NETA. TThe overall number of participants analyzed represents the number of participants evaluable at that time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 235 | 204 | 233
score on a scale | -3.9 (0.15) | -3.6 (0.16) | -3.6 (0.15)

15. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean Overall Pelvic Pain NRS Score At Week 104
Description: as for outcome 14
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 112 | 124
score on a scale | -4.2 (0.16) | -3.9 (0.17) | -4.0 (0.16)

16. Secondary Outcome: Percentage Of Participants Not Using Opioids For Endometriosis-associated Pain At Week 104
Description: Assessed based on usage of study-specified opioids for endometriosis-associated pain recorded daily in an electronic diary. Participants received protocol-specified opioids for treatment of endometriosis-associated pain as needed for pain but not prophylactically.
Time Frame: Week 104
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 277 | 247 | 275
percentage of participants | 91.0 [87.0 to 94.1] | 88.3 [83.6 to 92.0] | 90.5 [86.5 to 93.7]

17. Secondary Outcome: Percentage Of Participants Not Using Analgesics For Endometriosis-associated Pain At Week 104
Description: Assessed based on usage of study-specified analgesics for endometriosis-associated pain recorded daily in an electronic diary. Participants received protocol-specified analgesics for treatment of endometriosis-associated pain as needed for pain but not prophylactically.
Time Frame: Week 104
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 277 | 247 | 275
percentage of participants | 75.1 [69.6 to 80.1] | 76.5 [70.7 to 81.7] | 76.0 [70.5 to 80.9]

18. Secondary Outcome: Percentage Of Participants Who Are "Better" Or "Much Better" On The PGIC For NMPP At Week 52
Description: The PGIC for NMPP is a 1-item questionnaire designed to assess participant's impression of change in the severity of pain when they are not menstruating. The questionnaire used a 7-point response scale: much better, better, a little better, the same, a little worse, worse, or much worse.
Time Frame: Week 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 221 | 202 | 230
percentage of participants | 85.5 [80.18 to 89.88] | 86.1 [80.59 to 90.59] | 79.1 [73.30 to 84.19]

19. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean Dyspareunia NRS Scores At Week 52
Description: Assessed using an NRS score (11-point scale) for pain recorded daily in an electronic diary. Participants were to report whether they had vaginal sexual intercourse and rated their level of pelvic pain during intercourse on a scale from 0 to 10, with 0 indicating no pain and 10 indicating pain as bad as you can imagine. The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 151 | 126 | 140
score on a scale | -3.3 (0.18) | -3.0 (0.19) | -3.0 (0.18)

20. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean Dyspareunia NRS Scores At Week 104
Description: as for outcome 19
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 79 | 61 | 69
score on a scale | -3.5 (0.21) | -2.9 (0.22) | -3.4 (0.21)

21. Secondary Outcome: Percentage Of Participants Who Are "Better" Or "Much Better" On The PGIC For Dyspareunia At Week 52
Description: The PGIC for dyspareunia is a 1-item questionnaire designed to assess participant's impression of change in the severity of their pain during sexual intercourse. The questionnaire used a 7-point response scale: much better, better, a little better, the same, a little worse, worse, or much worse.
Time Frame: Week 52
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 210 | 194 | 210
percentage of participants | 61.0 [54.00 to 67.59] | 61.9 [54.62 to 68.72] | 60.0 [53.03 to 66.68]

22. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean Dyspareunia Functional Impairment At Week 52
Description: Assessed using the participant-modified Biberoglu and Behrman 5-point scale for dyspareunia recorded daily in an electronic diary. Participants were to report their pain during intercourse daily using the following response options: Severe (avoids intercourse because of pain), Moderate (intercourse painful to the point of causing interruption), Mild (tolerated pain), No pain (no pain during intercourse), or No intercourse (no intercourse for other reasons). Participants gave a possible score of 0 (no pain) to 3 (severe). The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 174 | 143 | 160
score on a scale | -0.9 (0.06) | -0.9 (0.06) | -0.8 (0.06)

23. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In The Mean Dyspareunia Functional Impairment At Week 104
Description: as for outcome 22
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 90 | 68 | 73
score on a scale | -1.0 (0.06) | -0.9 (0.07) | -1.0 (0.07)

24. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In Severity Scores On The Patient Global Assessment (PGA) For Overall Pelvic Pain At Week 52
Description: The PGA for pelvic pain severity is a 1-item questionnaire designed to assess participant's impression of the severity of their pain. The questionnaire used a 5-point response scale; each response was given a numerical score: absent (0), mild (1), moderate (2), severe (3), or very severe (4). The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 232 | 206 | 226
score on a scale | -1.3 (0.06) | -1.2 (0.06) | -1.2 (0.06)

25. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In Severity Scores On The Patient Global Assessment (PGA) For Overall Pelvic Pain At Week 104
Description: as for outcome 24
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 159 | 146 | 168
score on a scale | -1.4 (0.07) | -1.4 (0.07) | -1.3 (0.07)

26. Secondary Outcome: Percentage Of Participants With Improvement, No Change, Or Worsening From Baseline In PGA Score For Overall Pelvic Pain At Week 52
Description: The PGA for pelvic pain severity is a 1-item questionnaire designed to assess participant's impression of the severity of their pain. The questionnaire used a 5-point response scale; each response was given a numerical score: absent (0), mild (1), moderate (2), severe (3), or very severe (4).
Time Frame: Week 52
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 232 | 206 | 226
percentage of participants
  Improvement (-1 to -4) | 81.5 | 69.9 | 72.6
  No Change (0) | 14.7 | 26.2 | 23.0
  Deterioration (+1 to +4) | 3.9 | 3.9 | 4.4

27. Secondary Outcome: Percentage Of Participants With Improvement, No Change, Or Worsening From Baseline In PGA Score For Overall Pelvic Pain At Week 104
Description: as for outcome 26
Time Frame: Week 104
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 159 | 146 | 168
percentage of participants
  Improvement (-1 to -4) | 85.5 | 82.2 | 80.4
  No Change (0) | 13.8 | 15.8 | 16.7
  Deterioration (+1 to +4) | 0.6 | 2.1 | 3.0

28. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In Function Impairment On The PGA For Function At Week 52
Description: The PGA for functional impairment is a 1-item questionnaire designed to assess participant's impression of how their pain affected their usual activities. The participants responded to the question: "How much were your daily activities limited by endometriosis over the last 4 weeks?" using a 5-point response scale; each response was given a numerical score: not at all (0), minimally (1), moderately (2), significantly (3), or very significantly (4). The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: Extension Study Population: all participants who enrolled into MVT-601-3103 study and received any amount of open-label study drug in MVT-601-3103 study. Study results are reported by pivotal study treatment, but all participants only received relugolix pus E2/NETA. The overall number of participants analyzed represents the number of participants evaluable at that time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 235 | 206 | 230
score on a scale | -1.6 (0.06) | -1.6 (0.06) | -1.6 (0.06)

29. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In Function Impairment On The PGA For Function At Week 104
Description: as for outcome 28
Time Frame: Week 104
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 164 | 150 | 170
score on a scale | -1.9 (0.07) | -1.9 (0.07) | -1.8 (0.07)

30. Secondary Outcome: Percentage Of Participants With Improvement, No Change, Or Worsening From Baseline In PGA Score For Function At Week 52
Description: The PGA for functional impairment is a 1-item questionnaire designed to assess participant's impression of how their pain affected their usual activities. The participants responded to the question: "How much were your daily activities limited by endometriosis over the last 4 weeks?" using a 5-point response scale; each response was given a numerical score: not at all (0), minimally (1), moderately (2), significantly (3), or very significantly (4).
Time Frame: Week 52
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 235 | 206 | 230
percentage of participants
  Improvement (-1 to -4) | 88.9 | 86.9 | 86.1
  No Change (0) | 8.1 | 12.6 | 10.0
  Deterioration (+1 to +4) | 3.0 | 0.5 | 3.9

31. Secondary Outcome: Percentage Of Participants With Improvement, No Change, Or Worsening From Baseline In PGA Score For Function At Week 104
Description: as for outcome 30
Time Frame: Week 104
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 164 | 150 | 170
percentage of participants
  Improvement (-1 to -4) | 92.7 | 92.0 | 91.2
  No Change (0) | 6.7 | 7.3 | 8.8
  Deterioration (+1 to +4) | 0.6 | 0.7 | 0

32. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In Each Of The Non-Pain EHP-30 Domains At Week 52
Description: Assessed using the following non-pain domains of the EHP-30 questionnaire: Control and Powerlessness (questions 12 through 17), Emotional Well-Being (questions 18 through 23), Social Support (questions 24 through 27), and Self-Image (questions 28 through 30). The score for each domain ranged from 0 to 100. Higher scores represent a greater impact of endometriosis. The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 232 | 207 | 229
score on a scale
  Control and Powerlessness | -43.7 (1.61) | -40.1 (1.66) | -39.5 (1.59)
  Emotional Well-being | -26.7 (1.51) | -24.4 (1.56) | -23.7 (1.49)
  Social Support | -28.8 (1.69) | -28.9 (1.74) | -28.7 (1.67)
  Self Image | -26.4 (1.70) | -23.1 (1.75) | -22.8 (1.68)

33. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In Each Of The Non-Pain EHP-30 Domains At Week 104
Description: as for outcome 32
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 167 | 151 | 173
score on a scale
  Control and Powerlessness | -47.5 (1.59) | -43.7 (1.63) | -41.9 (1.54)
  Emotional Well-being | -30.7 (1.60) | -26.5 (1.65) | -25.6 (1.56)
  Social Support | -33.2 (1.85) | -24.9 (1.90) | -29.7 (1.80)
  Self Image | -29.5 (1.88) | -25.8 (1.94) | -25.2 (1.83)

34. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In Dysmenorrhea Functional Impairment Score At Week 52
Description: Assessed using the participant-modified Biberoglu and Behrman 5-point scale for dysmenorrhea recorded daily in an electronic diary. Participants were to report their pain as related to functional impairment daily in an electronic diary using the following response options: Severe (in bed all day, incapacitation), Moderate (in bed part of the day, some loss of work efficiency), Mild (some loss of work efficiency), No pain (no pain associated with menstruation during past 24 hours), or did not menstruate during the past 24 hours. Participants gave a possible score of 0 (no pain) to 4 (did not menstruate). The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 235 | 204 | 233
score on a scale | -1.3 (0.04) | -1.3 (0.04) | -1.2 (0.04)

35. Secondary Outcome: Change From The Pivotal Phase 3 Study Baseline In Dysmenorrhea Functional Impairment Score At Week 104
Description: as for outcome 34
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 112 | 124
score on a scale | -1.3 (0.04) | -1.3 (0.05) | -1.2 (0.04)

36. Secondary Outcome: Change From Pivotal Phase 3 Study Baseline In NMPP Functional Impairment Score At Week 52
Description: Assessed using the participant-modified Biberoglu and Behrman 4-point scale for pelvic pain recorded daily in an electronic diary. Participants reported their pain daily in an electronic diary using the following response options: Severe (requires strong analgesics), Moderate (noticeable pelvic pain), Mild (occasional pelvic pain), or No pain (no pain during past 24 hours). Participants gave a possible score of 0 (no pain) to 3 (severe). The LS mean was presented by pivotal study treatment group and by visit.
Time Frame: Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 235 | 204 | 233
score on a scale | -1.0 (0.04) | -1.0 (0.05) | -1.0 (0.04)

37. Secondary Outcome: Change From Pivotal Phase 3 Study Baseline In NMPP Functional Impairment Score At Week 104
Description: as for outcome 36
Time Frame: Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 129 | 112 | 124
score on a scale | -1.2 (0.05) | -1.1 (0.05) | -1.1 (0.05)

38. Secondary Outcome: Percent Change From The Pivotal Phase 3 Study Baseline In BMD At Lumbar Spine (L1-L4), Femoral Neck, And Total Hip At Week 52
Description: Assessed by dual-energy X-ray absorptiometry (DXA) scan at lumbar spine, total hip, and femoral neck (same leg for each participant) at each designated time point. All participants who completed treatment or terminated from the study early were required to return for a 6-month post-treatment follow-up (PTFU) and a 12-month PTFU DXA scan (except if participant was beyond 14 months from last day on treatment). Participants were also to have clinical laboratory evaluations (vitamin D, thyroid stimulating hormone, parathyroid hormone, creatinine, calcium, and phosphorous) at the 6-month and 12-month PTFU only if the PTFU DXA scans showed a bone loss of ≥3% at the lumbar spine and/or total hip compared with the parent study baseline.
Time Frame: Week 52
Population: Extension Safety Population: all enrolled participants who received any amount of open-label study drug in MVT-601-3103. Study results are reported by pivotal study treatment, but all participants only received relugolix plus E2/NETA. The number analyzed represents the proportion of the overall number of participants analyzed with values at that time point.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 233 | 205 | 232
percent change
  Lumbar Spine (L1-L4): number analyzed (Participants) | 233 | 204 | 232
  Lumbar Spine (L1-L4) | -0.69 (0.241) | -1.09 (0.256) | -0.09 (0.244)
  Femoral Neck: number analyzed (Participants) | 233 | 205 | 231
  Femoral Neck | -0.21 (0.277) | -0.84 (0.294) | 0.06 (0.280)
  Total Hip: number analyzed (Participants) | 233 | 205 | 231
  Total Hip | -0.10 (0.207) | -0.52 (0.219) | 0.27 (0.210)

39. Secondary Outcome: Percent Change From The Pivotal Phase 3 Study Baseline In BMD At Lumbar Spine (L1-L4), Femoral Neck, And Total Hip At Week 104
Description: as for outcome 38
Time Frame: Week 104
Population: Extension Safety Population: all enrolled participants who received any amount of open-label study drug in MVT-601-3103. Study results are reported by pivotal study treatment, but all participants only received relugolix plus E2/NETA. The overall number of participants analyzed represents the number of participants evaluable at that time point.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Relugolix Plus Delayed E2/NETA (Group B): Relugolix 40 mg monotherapy (once daily) for 12 weeks, followed by oral relugolix 40 mg once daily coadministered with E2 (1mg) and NETA (0.5 mg) for 12 weeks in the pivotal study and Relugolix 40 mg once daily co-administered with E2/NETA for 80 weeks in this extension study.
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 163 | 150 | 173
percent change
  Lumbar Spine (L1-L4) | -0.45 (0.295) | -0.56 (0.310) | -0.09 (0.292)
  Femoral Neck: number analyzed (Participants) | 163 | 150 | 170
  Femoral Neck | 0.24 (0.325) | -0.44 (0.341) | -0.05 (0.324)
  Total Hip: number analyzed (Participants) | 163 | 150 | 170
  Total Hip | 0.82 (0.268) | 0.10 (0.281) | 0.69 (0.267)

40. Secondary Outcome: Change From Pivotal Phase 3 Study Baseline In Predose Serum Concentrations Of Estradiol At Week 52
Description: Blood samples were collected from participants for estradiol measurements at each specified timepoints. Estradiol concentrations were measured using an immuno-enzymatic assay based on a commercially available kit.
Time Frame: Week 52
Population: Extension Safety Population: all enrolled participants who received any amount of open-label study drug in MVT-601-3103. Study results are reported by pivotal study treatment, but all participants only received relugolix Plus E2/NETA. The number of participants analyzed represents the proportion of the participants with values at that time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 210 | 185 | 201
pg/mL | -55.22 (99.636) | -77.76 (125.791) | -62.07 (90.031)

41. Secondary Outcome: Change From Pivotal Phase 3 Study Baseline In Predose Serum Concentrations Of Estradiol At Week 104
Description: as for outcome 40
Time Frame: Week 104
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
Number analyzed (Participants) | 148 | 133 | 157
pg/mL | -51.72 (106.801) | -74.68 (138.840) | -64.39 (104.463)

ADVERSE EVENTS:
Time Frame: Week 24/Baseline up to Week 104
Description: Extension Safety Population: all enrolled participants who received any amount of open-label study drug in MVT-601-3103. Study results are reported by pivotal study treatment, but all participants only received relugolix Plus E2/NETA.
Arm/Group | Relugolix Plus E2/NETA (Group A) | Relugolix Plus Delayed E2/NETA (Group B) | Placebo (Group C)
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/247 | 0/275
Serious Adverse Events (participants affected / at risk) | 7/277 | 19/247 | 18/275
Other Adverse Events (participants affected / at risk) | 173/277 | 106/247 | 151/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix Plus E2/NETA (Group A) (N=277) | Relugolix Plus Delayed E2/NETA (Group B) (N=247) | Placebo (Group C) (N=275)
Goitre (Endocrine disorders) | 0 | 0 | 2
Eye pain (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 2 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Personality disorder (Psychiatric disorders) | 1 | 0 | 0
Suicide threat (Psychiatric disorders) | 1 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Borderline personality disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 1 | 0
Panic disorder (Psychiatric disorders) | 0 | 0 | 1
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 3 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Broad ligament tear (Reproductive system and breast disorders) | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 2
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relugolix Plus E2/NETA (Group A) (N=277) | Relugolix Plus Delayed E2/NETA (Group B) (N=247) | Placebo (Group C) (N=275)
Headache (Nervous system disorders) | 38 | 18 | 38
Vulvovaginal mycotic infection (Infections and infestations) | 28 | 12 | 15
Nasopharyngitis (Infections and infestations) | 24 | 14 | 22
Vaginal infection (Infections and infestations) | 22 | 18 | 17
Urinary tract infection (Infections and infestations) | 18 | 12 | 14
Depressed mood (Psychiatric disorders) | 15 | 7 | 15
Vulvovaginal dryness (Reproductive system and breast disorders) | 15 | 7 | 9
Corona virus infection (Infections and infestations) | 13 | 18 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT03654274/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT03654274/SAP_001.pdf